CLINICAL TRIAL: NCT02455427
Title: Safety of Transcranial Direct Current Stimulation in the Subacute Phase After Stroke
Acronym: NEUROSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 225014
Record Dates: First submitted 2015-04-24; First posted 2015-05-27 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: transcranial direct current stimulation; conventional physical therapy
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS+ Physical Therapy (Active Comparator): Active tDCS (transcranial direct current stimulation) will be applied for 20 minutes. After active session of tDCS, the patient will receive physical therapy for 60 minutes. Number of treatment sessions: 6 (3 times a week, for 2 weeks)
  Interventions: Device: Active tDCS; Other: Physical Therapy
- Sham tDCS+Physical Therapy (Sham Comparator): Sham tDCS (transcranial direct current stimulation) will be applied for 20 minutes. After sham session of tDCS, the patient will receive physical therapy for 60 minutes.
  Number of treatment sessions: 6 (3 times a week, for 2 weeks)
  Interventions: Other: Physical Therapy; Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active tDCS will be applied with the anode positioned over the ipsilesional primary motor cortex and the cathode over the contralateral supraorbital region for 20 minutes (1mA).
  Arms: Active tDCS+ Physical Therapy
Other: Physical Therapy — Physical therapy will be administered for 60 minutes
Device: Sham tDCS — In sham tDCS, no current will be delivered through the tDCS device.
  Arms: Sham tDCS+Physical Therapy

SUMMARY:
Stroke is the second cause of death worldwide and represented the first cause of death in Brazil between 2006 and 2010. Most patients survive, and there is a need to develop cost-effective rehabilitation strategies to decrease the burden of disability from stroke.

This study addresses this important issue, by evaluating, in the early phase post-stroke, effects of motor conventional physical therapy associated or not with transcranial direct current stimulation (tDCS).

DETAILED DESCRIPTION:
The investigators main goal is to confirm the safety of transcranial direct current stimulation (tDCS) associated with conventional physical therapy, compared to conventional physical therapy associated with sham tDCS, for upper limb rehabilitation in an early phase (72 hours until 6 weeks) after stroke. Patients will be randomized to receive one of these two treatments, 3 times per week, for 2 weeks. Adverse effects will be monitored during each session. The working hypothesis is that conventional physical therapy associated with active tDCS in the subacute phase of ischemic stroke will be as safe as conventional therapy alone. The investigators will also preliminarily evaluate the efficacy of active tDCS associated with conventional therapy, compared to conventional therapy alone, in improvement of upper limb motor impairment. The investigators secondary goals are: 1) To compare effects of the above mentioned interventions on disability, spasticity and quality of life, in patients at an early stage after stroke ( subacute phase), immediately after treatment and 3 months later. The investigators hypothesis is that the association of conventional physical therapy and active tDCS will lead to better outcomes than conventional therapy alone. Patients will be assessed before the first session and after the last session of treatment, as well as 3 months after the last session of treatment.

Preliminary data about structural and functional connectivity will be collected in order to plan future studies related to mechanisms of tDCS in the subacute phase after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke confirmed by computed tomography or magnetic resonance imaging, with onset between 72 hours and 6 weeks before enrollment.
* Unilateral paresis of upper limb
* National Institute of Health Stroke Scale ( NIHSS) score of at least 1 point in items 5a or 5b .
* Ability to provide written informed consent (patient ou legal representative).

Exclusion Criteria:

* Lesions affecting the corticomotor pathway in the hemisphere contralateral to the stroke.
* Neurologic diseases except migraine.
* Modified Rankin Scale > 2 prior to stroke.
* Advanced systemic disease such as cancer or advanced chronic renal disease.
* Clinical instability such as uncontrolled cardiac arrhythmia or heart failure.
* Contraindication for physical therapy.
* Pregnancy.
* Absolute or relative contraindications to tDCS: metallic prosthesis in the head or neck; lesions on the scalp, history of neurosurgery, pacemaker.
* Comprehension aphasia
* Dementia
* Cerebellar stroke or ataxia caused by involvement of cerebellar pathways in the brainstem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Safety of the intervention as assessed by frequency of adverse events | 2 weeks
  frequency of adverse events in the active and sham arms

SECONDARY OUTCOMES:
Improvement post treatment as measured by the Modified Rankin Scale | 2 weeks and 14 weeks
  Improvement post treatment
Improvement post treatment as measured by the NIH Stroke Scale | 2 weeks and 14 weeks
  Improvement post treatment
Improvement post treatment as measured by the Stroke Impact Scale | 2 weeks and 14 weeks
  Improvement post treatment
Upper limb subscale of Fugl Meyer Assessment of Sensorimotor recovery after stroke | 2 weeks and 14 weeks
  Improvement post treatment
Improvement post treatment as measured by the Modified Ashworth Scale | 2 weeks and 14 weeks
  Improvement post treatment
Improvement post treatment as measured by the Motor Activity Log | 2 weeks and 14 weeks
  Improvement post treatment
Montreal Cognitive Assessment Test | 2 weeks and 14 weeks
  No cognitive deterioration post treatment
Structural Connectivity as measured by diffusion tensor imaging analysis | 2 weeks
  Improvement post treatment
Functional Connectivity as measured by resting-state functional magnetic imaging analysis | 2 weeks
  Improvement post treatment
Improvement post treatment as measured by the Barthel index | 2 week and 14 weeks
  Improvement post treatment
Safety of the intervention as assessed by frequency of adverse events | 14 weeks
  frequency of adverse events in the active and sham arms
Improvement post treatment as measured by Pittsburgh Sleep Quality Index | 2 week and 14 weeks
  Improvement post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Adriana B Conforto, MD Phd, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Danielle Boasquevisque, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Deidentified imaging data will be shared with collaborators

REFERENCES:
- [Derived] Takahashi MTC, Balardin JB, Bazan PR, Boasquevisque DS, Amaro Junior E, Conforto AB. Effect of transcranial direct current stimulation in the initial weeks post-stroke: a pilot randomized study. Einstein (Sao Paulo). 2024 Jun 24;22:eAO0450. doi: 10.31744/einstein_journal/2024AO0450. eCollection 2024. PMID 38922218
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411